CLINICAL TRIAL: NCT01933425
Title: Optimizing Surgical Conditions: Intraabdominal Distance During Gynecologic Laparoscopic Surgery With and Without Muscle Relaxation (The Measurement Study)
Brief Title: Optimizing Surgical Conditions During Gynecologic Laparoscopic Surgery With Deep Neuromuscular Blockade
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Matias Vested Madsen, research assistent, MD, Herlev Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NMBDK2013; 2013-001164-29 (EudraCT Number)
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Neuromuscular Blockade
Keywords: surgical conditions; laparoscopy
MeSH Terms: interventions — Rocuronium; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep neuromuscular block followed by no neuromuscular block (Active Comparator): Deep neuromuscular blockade (PTC 0-1) with rocuronium 1 mg/kg followed by no neuromuscular blockade with sugammadex 8 mg/kg and placebo reversal.
  Measurements of intraabdominal distance during deep neuromuscular blockade and without neuromuscular blockade
  Interventions: Drug: rocuronium; Drug: sugammadex; Drug: placebo
- No neuromuscular block followed by deep neuromuscular block (Placebo Comparator): No neuromuscular blockade with placebo followed by deep neuromuscular blockade (PTC 0-1) with rocuronium 1 mg/kg and reversal with sugammadex 8 mg/kg.
  Measurements of intraabdominal distance during no neuromuscular blockade and during deep neuromuscular blockade.
  Interventions: Drug: rocuronium; Drug: sugammadex; Drug: placebo

INTERVENTIONS:
Drug: rocuronium
Drug: sugammadex
Drug: placebo

SUMMARY:
To investigate if deep neuromuscular blockade improves intraabdominal volume compared to no neuromuscular blockade in patients scheduled for gynecologic laparoscopic surgery with pneumoperitoneum 12 mmHg.

Hypothesis:

Deep neuromuscular blockade improves intraabdominal space (the distance from promontorium to skin surface, cm) compared to no neuromuscular blockade.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years old
* elective laparoscopic operation
* can read and understand Danish
* informed consent

Exclusion Criteria:

* BMI > 30 kg/cm2
* known allergy to medications that are included in the project,
* severe renal disease, defined by S-creatinine> 0,200 mmol/L, GFR < 30ml/min or hemodialysis),
* neuromuscular disease that may interfere with neuromuscular data,
* lactating or pregnant,
* impaired liver function,
* converting to laparotomy,
* perioperative use of neuromuscular blocking agents before randomization,
* pneumoperitoneum set to >12 mmHg on the insufflator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matias Vested Madsen, MD, Principal Investigator — Department of Anesthesiology Herlev Hospital; Olav Istre, MD, DMSc, professor, Study Director — Department of minimal invasive gynecology, Aleris-Hamlet, Copenhagen
Locations (1):
- Department of minimal invasive gynecology Aleris-Hamlet Private Hospital, Copenhagen, Søborg, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Carried out between November 2013 and April 2014. Center for Minimal Invasive Gynaecology, Aleris-Hamlet Hospital Copenhagen, Denmark.
  A total of 25 patients were eligible in the study period, of which nine declined to participate, and two were excluded due to the fact that they did not speak Danish. All 14 patients completed the study
Groups:
- Deep Neuromuscular Block First Then no Neuromuscular Block: Deep neuromuscular blockade (PTC 0-1) with rocuronium 1 mg/kg followed by no neuromuscular blockade with sugammadex 8 mg/kg and placebo reversal.
  Measurements of intraabdominal distance during deep neuromuscular blockade and without neuromuscular blockade
  rocuronium
  sugammadex
  placebo
- No Neuromuscular Block First Then Deep Neuromuscular Block: No neuromuscular blockade with placebo followed by deep neuromuscular blockade (PTC 0-1) with rocuronium 1 mg/kg and reversal with sugammadex 8 mg/kg.
  Measurements of intraabdominal distance during no neuromuscular blockade and during deep neuromuscular blockade.
  rocuronium
  sugammadex
  placebo
Period: Overall Study
Arm/Group | Deep Neuromuscular Block First Then no Neuromuscular Block | No Neuromuscular Block First Then Deep Neuromuscular Block
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Females
Arm/Group | Patient Characteristics in 14 Women
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
BMI [Mean (Standard Deviation); unit: kg/m2] | 22.2 (2.6)
Number of patients with previous abdominal surgery [Number; unit: participants] | 7
Number of patients with 0 pregnancies [Number; unit: participants] | 6
Number of patients with 1 pregnancy [Number; unit: participants] | 3
Number of patients with 2 pregnancies [Number; unit: participants] | 2
Number of patients with 3 pregnancies [Number; unit: participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Intraabdominal Distance (Centimeters)
Description: Difference in intraabdominal distance from promontorium to the edge of the trocar in umbilicus at 12 mmHg with and without deep neuromuscular blockade (PTC 0-1).
Time Frame: 1 hour
Population: Comparisons of changes in distances were performed with paired t-test.
Measure: Median (Full Range); unit: centimeters
Groups:
- Deep Neuromuscular Block: Intraabdominal distance during deep neuromuscular blockade (PTC 0-1).
- No Neuromuscular Block: Intraabdominal distance during no neuromuscular block
Arm/Group | Deep Neuromuscular Block | No Neuromuscular Block
Number analyzed (Participants) | 14 | 14
centimeters | 9.3 [8.6 to 9.6] | 9.0 [8.2 to 9.5]
Statistical Analysis 1: Comparison: Deep Neuromuscular Block vs No Neuromuscular Block; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [0.07 to 0.59]

2. Secondary Outcome: Intraabdominal Distance (Centimeters)
Description: Difference in intraabdominal distance from promontorium to the edge of the trocar in umbilicus at 8 mmHg with and without deep neuromuscular blockade (PTC 0-1).
Time Frame: 1 hour
Population: Comparisons of changes in distances were performed with paired t-test
Measure: Median (95% Confidence Interval); unit: centimeters
Arm/Group | Deep Neuromuscular Block | No Neuromuscular Block
Number analyzed (Participants) | 14 | 14
centimeters | 8.6 [7.7 to 8.9] | 8.2 [7.4 to 8.8]
Statistical Analysis 1: Comparison: Deep Neuromuscular Block vs No Neuromuscular Block; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 0.3, 95% CI 2-sided [0.06 to 0.54]

3. Secondary Outcome: Surgical Conditions During Suturing of the Abdominal Fascia
Description: Optimal (score 1) Good (score 2) Acceptable (score 3) Poor (score 4)
Time Frame: 1 hour
Population: Evaluation of surgical conditions was compared using Mann-Whitney U-test.
Measure: Number; unit: participants
Groups:
- Deep Neuromuscular Blockade: Deep neuromuscular blockade (PTC 0-1) with rocuronium 1 mg/kg followed by no neuromuscular blockade with sugammadex 8 mg/kg and placebo reversal.
  Measurements of intraabdominal distance during deep neuromuscular blockade and without neuromuscular blockade
  rocuronium
  sugammadex
  placebo
- no Neuromuscular Blockade: No neuromuscular blockade with placebo followed by deep neuromuscular blockade (PTC 0-1) with rocuronium 1 mg/kg and reversal with sugammadex 8 mg/kg.
  Measurements of intraabdominal distance during no neuromuscular blockade and during deep neuromuscular blockade.
  rocuronium
  sugammadex
  placebo
Arm/Group | Deep Neuromuscular Blockade | no Neuromuscular Blockade
Number analyzed (Participants) | 7 | 7
participants
  Optimal (score 1) | 7 | 2
  Good (score 2) | 0 | 5
  Acceptable (score 3) | 0 | 0
  Poor (score 4) | 0 | 0

ADVERSE EVENTS:
Groups:
- Deep Neuromuscular Block First Then no Neuromuscular Block; No Neuromuscular Block First Then Deep Neuromuscular Block: Difference in intraabdominal distance comparing deep neuromuscular blockade (PTC 0-1) with no neuromuscular blockade.
Arm/Group | Deep Neuromuscular Block First Then no Neuromuscular Block | No Neuromuscular Block First Then Deep Neuromuscular Block
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes